CLINICAL TRIAL: NCT06736925
Title: Mechanistic Investigation of Omega-3 Fatty Acids Pretreatment Effects on Subconcussive Brain Injury
Brief Title: Omega-3 Fatty Acids and Subconcussive Head Impacts
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Keisuke Kawata, Associate Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 21334; R01NS137276 (NIH)
Record Dates: First submitted 2024-10-22; First posted 2024-12-17 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Subconcussive Head Impact; Omega-3 Fatty Acids
Keywords: Subconcussive brain injury; TBI; Soccer heading; Omega-3 fatty acids
MeSH Terms: interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Intervention Model Description: One group will be randomly assigned to take DHA+EPA, while the other group will be randomly assigned to take the placebo, organic soybean oil. Both groups will received identical stimuli of 20 soccer headings per session for a total of 2 sessions.
Who Masked: Participant, Investigator
Masking Description: Several co-investigators and undergraduate researchers will remain masked throughout the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo: Organic soybean oil pills (Placebo Comparator): We will use organic soybean oil pills ) as a placebo condition for the DHA+EPA group. One capsule contains 485 mg of organic soybean oil, including negligible amounts of DHA (1.1 mg), EPA (1.7 mg), and vitamin E (10 mg). Participants will ingest 5 capsules daily. Soybean oil is one of the most widely used vegetable oils in the world. Soybean oil contains polyunsaturated fats and 18-carbon omega-3 FA (total omega-3 FA of 73.9 mg per capsule), but very low levels of DHA and EPA, which makes it an excellent placebo counterpart when evaluating the effects of DHA/EPA. The placebo capsule's shelf life, composition, shape, size as the DHA+EPA active comparator.
  Interventions: Dietary Supplement: Organic soybean oil; Other: Soccer Heading Model
- Omega-3 Fatty Acids (EPA plus DHA) (Active Comparator): DHA+EPA capsules contain purified deep-sea fish oil, made from 100% wild-caught sardines and anchovies with a 3-year shelf life. The capsule shell is made from bovine limed bone with a size of 20 oblongs. Each soft gel capsule contains 480 mg of DHA, 205 mg of EPA, 145 mg of other omega-3 FA, and 10 mg of vitamin E. Participants in the DHA+EPA group will ingest 5 capsules daily [a total of 3.4 g/d: DHA (2.4 g), EPA (1.0 g)].
  Interventions: Dietary Supplement: Omega-3 Fatty Acids (EPA plus DHA); Other: Soccer Heading Model

INTERVENTIONS:
Dietary Supplement: Omega-3 Fatty Acids (EPA plus DHA) — DHA+EPA capsules contain purified deep-sea fish oil, made from 100% wild-caught sardines and anchovies with a 3-year shelf life. The capsule shell is made from bovine limed bone with a size of 20 oblongs. Each soft gel capsule contains 480 mg of DHA, 205 mg of EPA, 145 mg of other omega-3 FA, and 10 mg of vitamin E. Participants in the DHA+EPA group will ingest 5 capsules daily [a total of 3.4 g/d: DHA (2.4 g), EPA (1.0 g)].
  Arms: Omega-3 Fatty Acids (EPA plus DHA)
Dietary Supplement: Organic soybean oil — We will use organic soybean oil pills ) as a placebo condition for the DHA+EPA group. One capsule contains 485 mg of organic soybean oil, including negligible amounts of DHA (1.1 mg), EPA (1.7 mg), and vitamin E (10 mg). Participants will ingest 5 capsules daily. Soybean oil is one of the most widely used vegetable oils in the world. Soybean oil contains polyunsaturated fats and 18-carbon omega-3 FA (total omega-3 FA of 73.9 mg per capsule), but very low levels of DHA and EPA, which makes it an excellent placebo counterpart when evaluating the effects of DHA/EPA. The placebo capsule's shelf life, composition, shape, size as the DHA+EPA active comparator.
  Arms: Placebo: Organic soybean oil pills
Other: Soccer Heading Model — A standardized and reliable soccer heading protocol will be used for the experiment. A triaxial accelerometer (G-force tracker) embedded in a head-band pocket and positioned directly below the external occipital protuberance (inion) to monitor linear and rotational head accelerations. A JUGS soccer machine will be used to simulate a soccer throw-in with a standardized ball speed of 30 mph. The ball speed is similar to when soccer players make a long throw-in from the sideline to mid-field. Soccer players frequently perform this maneuver during practice and games. Subjects will stand approximately 40ft away from the machine to perform the heading. Participants perform 20 headers with 1 header per 30 seconds. The subjects will be instructed to direct the ball back toward the JUGS soccer machine in the air.

SUMMARY:
The purpose of the proposed double-blind, randomized placebo-controlled trial is to understand how supplementation with fish oil [docosahexaenoic acid (DHA) and eicosapentaenoic acid (EPA)] promote brain health against soccer heading. The study involves taking DHA+EPA or placebo, questionnaires, blood draws, brain imaging, tests to evaluate heart function, and soccer headings.

DETAILED DESCRIPTION:
The purpose of the proposed study is to determine whether, and to what extent, supplementation with omega-3 fatty acids [docosahexaenoic acid (DHA) and eicosapentaenoic acid (EPA)] can maintain or promote neural wellbeing against repetitive subconcussive head impacts. This study will also characterize what aspects of brain cellular and physiologic resiliencies are enhanced by supplementation in adult soccer players (aged 18-30 years old). A sub-cohort of participants who meet criteria for ADHD diagnosis will be part of exploratory analysises.

ELIGIBILITY:
Inclusion Criteria:

* Between age 18-30
* Current or former soccer player
* At least 5 years of soccer heading experience
* Have internet access
* Willing to commit to avoid any sport activity that purposefully uses one's head to maneuver during the study period (American football, ice-hockey, rugby, wrestling, and soccer heading).

Exclusion Criteria:

* Any head or neck injury within 6 months before the study
* Implanted metal/magnetic devices (e.g., orthodontic braces
* Diagnosed autonomic or cardiovascular diseases (e.g., hypertension)
* Consuming oily fish (2 servings or more/month: salmon, bluefin, swordfish, anchovies)
* Allergy to fish or shellfish
* Consuming omega-3 FA supplements including plant-based (e.g., flaxseed) in the past 3 months.
* Pregnancy

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 208 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Blood Biomarkers | Baseline, 24 hours following 1st and 2nd heading sessions, 7 days following the 2nd heading session
  The primary outcome analyses will be comparing group differences (group x time interactions) in blood biomarkers, specifically NF-L (neurofilament light, ), tau (picogram per milliliter), GFAP (glial fibrillary acidic protein; nanograms per milliliter), UCH-L1 (ubiquitin C-terminal hydrolase-L1; picograms per milliliter), and S100B (S100 calcium binding protein B; nanograms per milliliter). The aggregation of all blood biomarkers will provide a comprehensive overview of the biofluid profile of the participant following repetitive head injury.
Diffusion Tensor Imaging | Baseline, 24 hours following 1st and 2nd heading sessions, 7 days following the 2nd heading session
  DTI will be used to derive mean diffusivity (MD; square millimeters per second) and fractional anisotropy (FA; a unitless value that ranges from 0 to 1, 0 = Isotropic, 1= Anisotropic) as indicators joint of axonal integrity (axonal microstructure) and connectivity of white matter tracts by measuring how water molecules move through brain tissues .
Sympathetic Reactivity | Baseline, 24 hours following 1st and 2nd heading sessions, 7 days following the 2nd heading session
  Sympathetic Reactivity will be measured by the Cold Pressor Test (CPT). CPT is a general assessment of the ability of the sympathetic nervous system to become activated. The main metric will be changes in mean arterial pressure (MAP) following soccer headings. This test will be performed by submerging a participants hand into cold water for 2 minutes while autonomic and hemodynamic variables are recorded. At each data collection, participants will be instrumented for the measurement of heart rate (electrocardiogram) and continuous blood pressure. Participants will rest quietly for ~10 minutes before the CPT begins. The test takes 2 minutes.
Near Point Convergence | Baseline, 24 hours following 1st and 2nd heading sessions, 7 days following the 2nd heading session
  Using the accommodative ruler, a target (14-point letter) will be moved toward the eyes at a rate of 1-2 cm/s. NPC will be recorded when participants report diplopia has occurred, or the tester observes eye misalignment. The assessment will be repeated twice, and the mean near point convergence value will be used for analyses.
King-Devick test | Baseline, 24 hours following 1st and 2nd heading sessions, 7 days following the 2nd heading session
  The King-Devick test (KDT) consists of a total of 145 saccades while rapidly reading numbers aloud to complete the test. The KDT will be administered on a tablet. The total time (in seconds) will be used for analysis.

SECONDARY OUTCOMES:
Neurite Orientation Dispersion and Density Imaging (NODDI) | Baseline, 24 hours following 1st and 2nd heading sessions, 7 days following the 2nd heading session
  NODDI metrics will be derived from the the diffusion tensor images using the NODDI toolbox v1.0 in Matlab. Maps of neurite density (ND), orientation dispersion (OD), and intracellular volume fraction (ICVF) will be generated.
Resting-state functional connectivity | Baseline, 24 hours following 1st and 2nd heading sessions, 7 days following the 2nd heading session
  Resting-state connectivity will be examined throughout the whole brain and specific seeded regions including the dorsolateral prefrontal cortex (DLPFC), angular gyrus, and cingulate gyrus.
Cardiovagal baroreflex sensitivity | Baseline, 24 hours following 1st and 2nd heading sessions, 7 days following the 2nd heading session
  Spontaneous cardiovagal baroreflex sensitivity (cBRS) will be collected over the last 5 minutes before the CPT. Baroreflex sequences of 4 consecutive cardiac cycles will be captured using WinCPRS software, for which directional changes in the R-R interval and corresponding systolic blood pressure will be identified. Sequences will be detected when changes in systolic blood pressure are ≥1mmHg and the variation in R-R interval is ≥5miliseconds. Only sequences with an R2 ≥0.85 will be deemed acceptable. The mean of the regression slope will be calculated as the cBRS gain and used for analysis
Heart rate variability | Baseline, 24 hours following 1st and 2nd heading sessions, 7 days following the 2nd heading session
  Leading up to and during the cold pressor test (CPT) heart rate will be monitored via 3-lead ECG. Resting-state heart rate variability and spontaneous cardiovagal baroreflex sensitivity (cBRS) will be monitored over the last 5 minutes before the CPT. Using the R-R interval data collected from the ECG recordings during 5 minutes of paced breathing, time domain analyses will be performed to estimate overall heart rate variability and provide insight into cardiac parasympathetic activity.
Cognition | Baseline, 24 hours following 1st and 2nd heading sessions, 7 days following the 2nd heading session
  Cognitive function will be measured using the NIH Toolbox Cognition Battery, which has excellent reliability and validity to measure cognition in young adults, and has construct validity among those with TBI. Multiple forms will minimize learning effects. This battery examines 5 cognitive domains (executive function, episodic memory, language, working memory, and processing speed) and takes 20 minutes to complete on a tablet.
Cerebral Blood Flow | Baseline, 24 hours following 1st and 2nd heading sessions, 7 days following the 2nd heading session
  Perfusion imaging will be acquired to examine cerebral blood flow.
Metabolomics | Baseline, 24 hours following 1st and 2nd heading sessions, 7 days following the 2nd heading session
  Mitochondrial respiration related metabolites, including pyruvate, acetyl-CoA, citrate, isocitrate, alpha-ketogluterate, succinyl-CoA, succinate, fumarate, malate, and oxaloacetate will be assessed on blood samples. The aggregation of all metabolomic data will provide a comprehensive overview of the homeostasis of the participant following repetitive head injury.
Quantitative Susceptibility Mapping | Baseline, 24 hours following 1st and 2nd heading sessions, 7 days following the 2nd heading session
  Quantitative Susceptibility Mapping of whole brain, as well as regions of interest analysis, will be conducted to inspect the tissue and brain architectural response to head impacts and omega-3 fatty acid supplementation.

OTHER OUTCOMES:
Genetic markers | Baseline
  Several genetic markers that are known to associate with brain vulnerability will be assessed and regressed against our outcome measures. These genetic markers include, but not limited to, DARC, APOE, KIAA0319, BDNF, TPH2, COMT. Each marker will be compared to the other outcome measures to understand the full effect of the intervention on the genetic markers as a whole.
ADHD | Baseline
  Participants who meet criteria for ADHD diagnosis will be analyzed to address the interactive effects of DHA+EPA and head impacts in ADHD.

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University School of Public Health, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marchi N, Bazarian JJ, Puvenna V, Janigro M, Ghosh C, Zhong J, Zhu T, Blackman E, Stewart D, Ellis J, Butler R, Janigro D. Consequences of repeated blood-brain barrier disruption in football players. PLoS One. 2013;8(3):e56805. doi: 10.1371/journal.pone.0056805. Epub 2013 Mar 6. PMID 23483891
- [Background] Kawata K, Rubin LH, Takahagi M, Lee JH, Sim T, Szwanki V, Bellamy A, Tierney R, Langford D. Subconcussive Impact-Dependent Increase in Plasma S100beta Levels in Collegiate Football Players. J Neurotrauma. 2017 Jul 15;34(14):2254-2260. doi: 10.1089/neu.2016.4786. Epub 2017 Apr 27. PMID 28181857
- [Background] Puvenna V, Brennan C, Shaw G, Yang C, Marchi N, Bazarian JJ, Merchant-Borna K, Janigro D. Significance of ubiquitin carboxy-terminal hydrolase L1 elevations in athletes after sub-concussive head hits. PLoS One. 2014 May 7;9(5):e96296. doi: 10.1371/journal.pone.0096296. eCollection 2014. PMID 24806476
- [Background] Oliver JM, Jones MT, Kirk KM, Gable DA, Repshas JT, Johnson TA, Andreasson U, Norgren N, Blennow K, Zetterberg H. Serum Neurofilament Light in American Football Athletes over the Course of a Season. J Neurotrauma. 2016 Oct 1;33(19):1784-1789. doi: 10.1089/neu.2015.4295. Epub 2016 Mar 16. PMID 26700106
- [Background] Oliver JM, Anzalone AJ, Stone JD, Turner SM, Blueitt D, Garrison JC, Askow AT, Luedke JA, Jagim AR. Fluctuations in blood biomarkers of head trauma in NCAA football athletes over the course of a season. J Neurosurg. 2018 May 29;130(5):1655-1662. doi: 10.3171/2017.12.JNS172035. Print 2019 May 1. PMID 29807487
- [Background] Shahim P, Zetterberg H, Tegner Y, Blennow K. Serum neurofilament light as a biomarker for mild traumatic brain injury in contact sports. Neurology. 2017 May 9;88(19):1788-1794. doi: 10.1212/WNL.0000000000003912. Epub 2017 Apr 12. PMID 28404801
- [Background] Joseph JR, Swallow JS, Willsey K, Lapointe AP, Khalatbari S, Korley FK, Oppenlander ME, Park P, Szerlip NJ, Broglio SP. Elevated markers of brain injury as a result of clinically asymptomatic high-acceleration head impacts in high-school football athletes. J Neurosurg. 2018 Jul 3;130(5):1642-1648. doi: 10.3171/2017.12.JNS172386. Print 2019 May 1. PMID 29966462
- [Background] Tierney GJ, Higgins B. The incidence and mechanism of heading in European professional football players over three seasons. Scand J Med Sci Sports. 2021 Apr;31(4):875-883. doi: 10.1111/sms.13900. Epub 2021 Jan 18. PMID 33280186
- [Background] Peek K, Vella T, Meyer T, Beaudouin F, McKay M. The incidence and characteristics of purposeful heading in male and female youth football (soccer) within Australia. J Sci Med Sport. 2021 Jun;24(6):603-608. doi: 10.1016/j.jsams.2020.12.010. Epub 2020 Dec 26. PMID 33414022
- [Background] Russell ER, Mackay DF, Stewart K, MacLean JA, Pell JP, Stewart W. Association of Field Position and Career Length With Risk of Neurodegenerative Disease in Male Former Professional Soccer Players. JAMA Neurol. 2021 Sep 1;78(9):1057-1063. doi: 10.1001/jamaneurol.2021.2403. PMID 34338724
- [Background] Mackay DF, Russell ER, Stewart K, MacLean JA, Pell JP, Stewart W. Neurodegenerative Disease Mortality among Former Professional Soccer Players. N Engl J Med. 2019 Nov 7;381(19):1801-1808. doi: 10.1056/NEJMoa1908483. Epub 2019 Oct 21. PMID 31633894
- [Derived] Beauregard LH, Bazarian JJ, Johnson BD, Cheng H, Ellis G, Kronenberger W, Calder PC, Chen Z, Silveyra P, Quinn PD, Newman SD, Mickleborough TD, Kawata K. Investigating omega-3 fatty acids' neuroprotective effects in repetitive subconcussive neural injury: Study protocol for a randomized placebo-controlled trial. PLoS One. 2025 Apr 24;20(4):e0321808. doi: 10.1371/journal.pone.0321808. eCollection 2025. PMID 40273177